CLINICAL TRIAL: NCT04640922
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate Clinical Performance and Safety of the Gedea Pessary in Adult Women With Bacterial Vaginosis
Brief Title: Clinical Performance and Safety of the Gedea Pessary in Adult Women With Bacterial Vaginosis
Acronym: Nefertiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QRS-CL3-003; CIV-GB-20-09-034813 (Other: EUDAMED)
Record Dates: First submitted 2020-11-13; First posted 2020-11-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind placebo-controlled multi-centre study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gedea Pessary (Active Comparator): pHyph, vaginal tablet, daily in Part 1 and once weekly in Part 2
  Interventions: Device: Gedea Pessary pHyph
- Placebo (Placebo Comparator): placebo, vaginal tablet, daily in Part 1 and once weekly in Part 2
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Gedea Pessary pHyph — Vaginal tablet
  Arms: Gedea Pessary
Device: Placebo — Vaginal tablet
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind placebo-controlled multi-centre study to evaluate clinical performance, safety and local tolerability of initial and preventive treatment with Gedea Pessary in adult women with confirmed BV.

The study population will consist of post-menarchal, pre-menopausal females 18 years or older seeking for BV symptoms (fishy smell, irritation and burning).

Patients will be recruited at study sites' gynaecological and sexual health clinics and a total of 150 patients are planned to be randomised in the study.

On Day 0, patients will have gynaecological examination, vaginal samples taken, and will be randomised in a 4:1 relation to receive treatment with 6 doses of the Gedea Pessary or a vehicle control (placebo) to be self-administered daily (Days 0 to 5). Patients will be re examined at Day 7 (+2 days) for clinical cure rate.

Patients that are clinically cured at Day 7 will continue to the second part of the study and will be randomised in a 1:1 relation to either Gedea Pessary or placebo treatment, to be self administered once a week for a duration of 126 days.

Patients not clinically cured at Day 7 will be offered rescue treatment (metronidazole) for 7 days. They will return at Day 14 for clinical assessment and sampling for microbiome and mycobiome analysis, and if cured they will be assessed for recurrence up to Day 128. Patients that are not cured at Day 14 will be discontinued from the study.

Patients that are clinically cured at Day 7 and continuing in Part 2 will be followed up until confirmed recurrence or Day 128 if no recurrence. Vaginal samples will be taken by self-swab on Days 35, 63 and 91, a visit to the clinic will be performed at Day 63 and telephone follow up will be done at Days 35 and 91. Vaginal samples will also be taken at the visit on the Day of potential recurrence and/or at Day 128 if no recurrence.

Vaginal samples will be used for confirming the diagnosis (Nugent score on Day 0 and Day 7) and sequencing analysis of the vaginal microbiome and mycobiome (Days 0, 7, 35, 63, 91 and Day of confirmed recurrence or Day 128 if no recurrence).

Patient follow-up as regards to patient questionnaire/usability, AEs and BV recurrence notification will be handled with a mobile phone application. In case of a suspected BV recurrence, the patient should return to the clinic for confirmation of BV diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, post-menarchal, pre-menopausal women aged 18 years or older.
2. Diagnosis of BV according to Amsel's criteria, defined as having at least 3 of the 4 criteria.
3. Having decisional capacity and providing written informed consent.
4. Negative urine pregnancy test at screening.
5. Refrain from using any intravaginal products (i.e. contraceptive creams, gels, foams, sponges, lubricants or tampons, etc.) until Day 7 and the following 24 hours after each treatment during weekly treatment.
6. Refrain from sexual intercourse or use a condom until Day 7.
7. Willing to use contraception (if heterosexual) for 128 days.
8. Signed informed consent and willing and able to comply with all study requirements.

Exclusion Criteria:

1. Patients with known or apparent signs of other infectious causes of vaginitis (e.g.

   vulvovaginal candidiasis, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex, or human papillomavirus) at screening.
2. Anticipated menstruation during the treatment period (Day 0 till Day 5).
3. Patients who are pregnant or breastfeeding.
4. Patients who are planning to conceive within the 128 days study duration.
5. Patients who were treated for BV within the past 14 days.
6. Patients who are currently receiving antibiotic therapy unrelated to BV or have received antibiotic therapy within the past 14 days.
7. Patients who have used pH-modifying vaginal products within the last 14 days.
8. Patients who have received an investigational drug in a clinical investigation within 30 days prior to screening.
9. Known/previous allergy or hypersensitivity to any product constituent.
10. Any medical condition that in the Investigator's judgments would make the patient unsuitable for inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate on Day 7 | Day 7
  o Defined as absence of all of the following 3 Amsel criteria:
  1. Thin, white, yellow, homogenous discharge;
  2. Clue cells on microscopy (more than 20% of epithelial cells);
  3. Release of fishy odour "i.e. a positive whiff test" when alkali (10% KOH solution) is added.

SECONDARY OUTCOMES:
Safety and local tolerability of Gedea Pessary - based on reported treatment-emergent AEs up until Day 7. | Day 7
  Part 1
Clinical cure rate on Day 7, defined as clinical cure according to primary endpoint and Nugent score <4, i.e. both criteria have to be fulfilled. | Day 7
  Part 1
Difference between Day 7 and Days 35, 63, 91, 128 and/or Day of possible recurrence confirmation (assessed by Amsel criteria), respectively, in the occurrence of anaerobic vaginal dysbiosis as assessed by analysis of the vaginal microbiome. | Day 35, 63, 91, and 128, respectively
  Part 2

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (2):
  - Hoftekliniken, Helsingborg
  - Curakliniken, Malmo
- United Kingdom (3):
  - Derbyshire Community Health Services NHS Foundation Trust, Derby
  - Northamptonshire Healthcare NHS Foundation Trust (NHFT), Northampton
  - Nottingham University Hospitals NHS Trust, Nottingham